CLINICAL TRIAL: NCT02483767
Title: Gonadotropin-Releasing Hormone Agonist for the Preservation of Ovarian Function During Chemotherapy in Premenopausal Breast Cancer
Acronym: POF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PUMCH-BC-ovarian suppression
Record Dates: First submitted 2015-06-09; First posted 2015-06-29 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
Keywords: Premenopausal Breast Cancer; Preservation of Ovarian Function; Gonadotropin-Releasing Hormone Agonist
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard chemotherapy with goserelin (Experimental): standard chemotherapy with the GnRH agonist goserelin
  Interventions: Drug: goserelin; Drug: standard chemotherapy
- standard chemotherapy without goserelin (Active Comparator): standard chemotherapy without goserelin
  Interventions: Drug: standard chemotherapy

INTERVENTIONS:
Drug: goserelin — Gonadotropin-Releasing Hormone Agonist
  Other Names: Gonadotropin-Releasing Hormone Agonist
  Arms: standard chemotherapy with goserelin
Drug: standard chemotherapy — (Anthracyclines/cyclophosphamide) followed by paclitaxel or doxetaxel; doxetaxel/cyclophosphamide; doxetaxel or paclitaxel/Anthracyclines; fluorouraci/Anthracyclines/cyclophosphamide followed by doxetaxel or paclitaxel; doxetaxel/Anthracyclines/cyclophosphamide; Anthracyclines/cyclophosphamide;
  Other Names: AC-P; TC; TA; TAC; FAC followed by T; AC

SUMMARY:
The study is a prospective randomized control clinical trial which is sponsored by the researchers. The purpose of this study is to determine the effectiveness of Gonadotropin-Releasing hormone agonist on ovarian function for premenopausal breast cancer patients during chemotherapy. The premenopausal breast cancer patients will be randomly (1:1) enrolled to receive standard chemotherapy with the GnRH agonist goserelin (goserelin group) or standard chemotherapy without goserelin (chemotherapy alone group). All patients are stratified according to age (<35years vs.36-44years), hormone receptor status (HR+ or ER+ vs.HR- and ER-), chemotherapy regimen(3-4 cycles vs.6-8 cycles, and cyclophosphamide-based vs.noncyclophosphamide).The follow-up time will be at least 2years. The ovarian failure, follicle-stimulating hormone, estradiol and anti-Mullerian hormone, pregnancy outcomes and disease-free and overall survival will be compared between two groups to evaluate the effectiveness of protect against ovarian failure.

ELIGIBILITY:
Inclusion Criteria:

* The patients signed the written informed consent.
* Histologically proven stage I, II, or III breast cancer
* Must be candidates for adjuvant or neoadjuvant chemotherapy,
* Must be premenopausal.
* Trastuzumab is permitted in patients with human epidermal growth factor receptor 2 (HER2) overexpressing tumors.

Exclusion Criteria:

* The patients were previous chemotherapy;
* Evidence of distant metastases;
* Other malignancies in the previous 5 years.
* The patients were using GnRHa, progesterone, stimulate ovulation drugs, oral contraceptives, aromatase inhibitors, intrauterine device with hormone, subcutaneous preparations contraceptive drugs such as hormone drugs and instruments during 3 month preceding the start of chemotherapy.
* Pregnancy or lactation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2015-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
ovarian failure | 2 years
  Ovarian failure is defined as amenorrhea for the preceding 6 months and follicle-stimulating hormone (FSH) and E2 levels in the post -menopausal range 2 year after the end of chemotherapy.

SECONDARY OUTCOMES:
Ovarian dysfunction | 1 year
  Ovarian dysfunction is defined as amenorrhea for the preceding 3 months and follicle-stimulating hormone (FSH) and E2 levels in the post -menopausal range 1 year or 2year after the end of chemotherapy.
Time to the resumption of menstrual activity | 2 year
  Time to the resumption of menstrual activity will be assessed at 3month，1 year and 2year after the end of chemotherapy.
pregnancy | 5 year
  whether pregnancy will be accessed at 1year, 2year, 3year, 4year, 5year after the end of chemotherapy
DFS OS | 5 year
  Disease free survival (DFS) and overall survival (OS) will be assessed at 5years after the end of chemotherapy.
FSH,E2,AMH | 2 year
  FSH, estradiol, and anti-Mullerian hormone (AMH) levels in the postmenopausal range will be assessed at 3month，1 year and 2year after the end of chemotherapy.